CLINICAL TRIAL: NCT04012346
Title: Modulation of Cognition and Brain Connectivity by Noninvasive Brain Stimulation in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease
Acronym: LUSTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NV16-31868A
Record Dates: First submitted 2019-06-28; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: MCI patients with real iTBS (Active Comparator): Patients will receive real iTBS in a week-long sessions.
  Interventions: Device: Transcranial magnetic stimulation
- Sham Comparator: MCI patients with sham iTBS (Sham Comparator): Patients will receive sham iTBS in a week-long sessions.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Transcranial magnetic stimulation device will be used. Short protocol iTBS will be applied.

SUMMARY:
Alzheimer's disease (AD) has a detrimental impact on cognitive functions. Based on pilot studies results in patients with neurodegenerative brain diseases the investigators aim for promoting the brain plasticity and improving cognition by noninvasive brain stimulation (NIBS) in healthy young, healthy aged and subjects with mild cognitive impairment due to AD. Mild cognitive impairment (MCI) is an intermediate stage between the expected cognitive decline of normal aging and the more-serious decline of dementia. Different new brain targets, cognitive tasks and stimulation protocols will be tested and optimized for specific subject groups. Design of a functional MRI (fMRI) - repetitive transcranial magnetic stimulation (rTMS) - fMRI study will enable us to explore and identify effect of age, presence of the disease and genetic risk factor (APOE4) on repetitive transcranial magnetic stimulation (rTMS)-induced changes in cognition and related brain connectivity/activations. The study results will improve our understanding of healthy and pathological brain aging and will provide novel information about the usefulness of NIBS in specific subject groups. These results will have an important impact on future non-pharmacological treatment strategies.

DETAILED DESCRIPTION:
Intensified intermittent theta-burst stimulation (iTBS) protocol will be applied in the MCI study group. A two-parallel-group, randomized, placebo controlled design will be used. Ten MCI subjects will be stimulated in a week-long therapeutical sessions. Other ten MCI subjects will be stimulated with the same protocol using sham stimulation. The investigators will study the change in subjects immediately after and again at a two-weeks follow-up visit after the end of the last stimulation session.

ELIGIBILITY:
Inclusion Criteria:

* amnestic single or multi-domain mild cognitive impairment patients in accordance with diagnostic criteria (Albert et al., 2011)

Exclusion Criteria:

psychiatric disorders, including major depression, major vascular lesions, and other brain pathologies detected by MRI that might present with cognitive decline

* a cardio pacemaker or any MRI-incompatible metal in the body
* epilepsy
* any diagnosed psychiatric disorder
* alcohol/drug abuse
* lack of cooperation
* presence of dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Visual-attention task accuracy and reaction times | On the beginning of the study, after completion of week stimulation a two weeks after completion of stimulation sessions.
  Stroop task will be presented in fMRI

SECONDARY OUTCOMES:
Resting state measurement | On the beginning of the study, after completion of week stimulation a two weeks after completion of stimulation sessions.
  The effect of stimulation on the resting state networks will be studied using fMRI measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Ceitec Masaryk University, Brno, Czechia